CLINICAL TRIAL: NCT05847543
Title: A Study to Develop, Evaluate, and Validate a Tool to Infer/Predict an Estimated Microbiome Profile
Brief Title: Building an AI to Infer/Predict an Estimated Stool Microbiome Profile
Acronym: Poobiome
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: KK Women's and Children's Hospital (Other Government); National University Hospital, Singapore (Other); University of Malaya (Other); Thammasat University Hospital (Other); Mount Elizabeth Medical Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: EBB19GC16961-A
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Microbiome; Artificial Intelligence; Stool
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-weaned Children: Children who have not started weaning food
  Interventions: Other: Stool diaper data and sample collection
- Weaned Children (Non-Caucasian): Non-Caucasian children who have started weaning food
  Interventions: Other: Stool diaper data and sample collection
- Weaned Children (Caucasian): Caucasian children who have started weaning food
  Interventions: Other: Stool diaper data and sample collection

INTERVENTIONS:
Other: Stool diaper data and sample collection — Stool diaper data and sample collection

SUMMARY:
This is a study to collect data to build, evaluate and validate (test) a tool to infer/predict an estimated microbiome (community of microorganisms such as bacteria, fungi and viruses that exists in a particular environment) profile. The study will take place at several hospitals/clinics across Singapore, Malaysia, and Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged from 0 to 18 months old
2. Parent(s) should have access to the internet and a smartphone or tablet to upload stool data and complete the study questionnaires in the OneBiome web-platform.
3. Parent(s) should be able to comprehend the content of the study and to complete the study procedures in English.
4. Written consent from parent.

Exclusion Criteria:

1. Parent(s) incapable of completing the study questionnaires and uploading of the stool data using smart phone or tablet with internet.
2. Children born before gestational age 37 weeks.
3. Any other family member is enrolled in the study
4. Incapability of parents of children to comply with study protocol or Investigator's uncertainty about the willingness or ability of the parents of children to comply with the protocol requirements.

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term children aged 0 to 18 months old
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
To collect stool data and stool samples for full microbiome analysis. To collect stool images, stool data and stool samples for full microbiome analysis | 7 days
  To collect stool data and stool samples for full microbiome analysis.
  To collect stool images, stool data and stool samples for full microbiome analysis

SECONDARY OUTCOMES:
To assess the microbiome composition in the stool sample of the subject | 7 days
  To assess the microbiome composition in the stool sample of the subject
To assess the dietary pattern based on Food Frequency Questionnaire (FFQ) | 7 days
  To determine/assess the eating/dietary pattern of the participants based on the Food Frequency Questionnaire (FFQ) data and reflect insights in the OneBiome report
To explore the association between microbiome composition and known factors that influence the microbiome in early life | 7 days
  To explore the association between microbiome composition and known factors that influence the microbiome in early life including mode of delivery, antibiotic prophylaxis, infant feeding patterns and diet

OTHER OUTCOMES:
The accuracy level of the stool AI in predicting the stool consistency using BITSS versus the scores provided by parents | 7 days
  The accuracy level of the stool AI in predicting the stool consistency using BITSS 4-point scale versus the scores provided by parents on the same 4-point scale

CONTACTS AND LOCATIONS:
Locations (4):
- University Malaya Medical Center, Kuala Lumpur, Malaysia
- Singapore (2):
  - Mount Elizabeth Medical Centre, Singapore
  - KK Women's and Children's Hospital, Singapore
- Thammasat University Hospital, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No